CLINICAL TRIAL: NCT06358820
Title: Exploring the Effectiveness and Safety of Amino Acid Peritoneal Dialysis Solution in Improving Nutritional Status in Maintenance Peritoneal Dialysis Patients: a Multicenter, Open, Prospective, Self Controlled Clinical Study
Brief Title: Exploring the Effectiveness and Safety of Amino Acid Peritoneal Dialysis Solution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The People's Hospital of Gaozhou (Other)
Responsible Party: Principal Investigator, deng shanshan, Researcher, The People's Hospital of Gaozhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHGaozhou
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Exploring the Effectiveness and Safety of Amino Acid Peritoneal Dialysis Solution
Keywords: amino acid peritoneal dialysis solution；peritoneal dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Control (Other): Compare the nutritional and safety indicators of the subjects before treatment and during the third and sixth months of treatment.
  Interventions: Drug: Amino acid peritoneal dialysis solution

INTERVENTIONS:
Drug: Amino acid peritoneal dialysis solution — Each subject received treatment with 1 bag of amino acid peritoneal dialysis daily and 2-4 bags of glucose peritoneal dialysis solution daily for 6 months

SUMMARY:
This study adopts a multicenter, open, prospective, and self controlled study design, in which each participant serves as their own control before and after receiving amino acid peritoneal dialysis solution treatment to compare changes in their nutritional status. Each subject received treatment with 1 bag of amino acid peritoneal dialysis per day and 2-4 bags of glucose peritoneal dialysis solution per day for 6 months (the amount of glucose peritoneal dialysis solution used was determined based on the treatment plan selected by the patient during the screening period when they entered the study).Before treatment and during the 3rd and 6th months of treatment, subjects were evaluated for various efficacy and safety indicators, and any adverse or serious adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. For uremic patients with malnutrition during the screening period, maintenance peritoneal dialysis should be performed for at least 3 months. The standard for malnutrition should meet at least two of the following items: (1) serum albumin level<3.5g/dL (35g/L), (2) prealbumin<300mg/L, (3) modifiedSubjective Global Assessment (SGA) with a score of>7;
2. Blood urea nitrogen ≤ 38mmol/L;
3. The patient's age is between 18 and 75 years old;
4. The patient signs an informed consent form.

Exclusion Criteria:

1. Individuals who are allergic to any amino acids or excipients in this product
2. More than one occurrence of peritonitis in the past three months; Peritonitis or hospitalization within the past month;
3. Patients with hyperthyroidism, systemic infection, fever, and other high catabolic metabolic diseases, as well as those who are taking drugs that affect tissue metabolism, such as corticosteroids;
4. Congenital amino acid metabolism deficiency disease, acute severe pancreatitis, severe hyperbilirubinemia 5. Patients with malignant tumor metastasis or spread, residual cancer after treatment, coagulation dysfunction, aplastic anemia, heart, brain, lung and other serious system diseases;

6. Possible kidney transplantation during the trial period; 7. Active phase of hepatitis B or C, liver cirrhosis, active liver disease, liver dysfunction, or positive serum reaction of human immunodeficiency virus (HIV); 8. Those who have participated in clinical trials of other drugs within the three months prior to enrollment; 9. Pregnant and lactating women; 10. Those who are mentally unable to cooperate; 11. Failure to sign a written informed consent form; 12. Unable or unwilling to comply with the experimental protocol approved by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gaozhou People's Hospital, Gaozhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng S, Xuan H, Chen L, Su X, Su Y, Lu Y, Zhu M, Yang X, Luo C, Shi W. Overnight-dwelled amino acid-based peritoneal dialysis solutions for malnutrition in CAPD: a prospective real-world study. Int Urol Nephrol. 2026 Feb;58(2):661-671. doi: 10.1007/s11255-025-04749-y. Epub 2025 Aug 27. PMID 40864356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self Control
Started | 149 (A total of 150 cases signed informed consent forms to participate in the clinical study, with 1 screening failure, resulting in 149 cases entering the clinical research.)
Completed | 128 (A total of 142 patients (95.3%) had at least one efficacy assessment.The withdrawal reasons included PD-related condition deterioration requiring treatment (n = 1, 4.76%), kidney transplantation (n = 3, 14.29%) , patient non-compliance with study protocol, serious adverse events (n = 11, 52.38%) and patient voluntary withdrawal (n = 6, 28.57%))
Not Completed | 21
Not completed — Adverse Event | 11
Not completed — kidney transplantation | 3
Not completed — patient voluntary withdrawal | 6
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Patients who completed one efficacy evaluation were defined as having completed the study.149 patients were enrolled, with 142 patients undergoing at least one efficacy evaluation.
Arm/Group | Enrolled
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  149: Female | 78
  149: Male | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 149
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 149
Duration of CAPD（Continuous ambulatory peritoneal dialysis） [Mean (Standard Deviation); unit: years] | 2.67 (1.16)
Residual urine [Median (Inter-Quartile Range); unit: ml/day] | 300 [50 to 650]

OUTCOME MEASURES:

1. Primary Outcome: Blood Albumin
Description: Changes in blood albumin levels
Time Frame: 6 months
Population: All included subjects received at least 1 dose of study treatment and had data for efficacy evaluation at at least 1 post-treatment observation time point.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Self Control
Number analyzed (Participants) | 142
g/L | 4.02 (3.64)
Statistical Analysis 1: Comparison: Self Control; Outcome Measure were assessed at baseline and every month during the 6-month study; Test type: Superiority — >0.15 g/dL change in albumin from baseline to month 6 was anticipated; p < 0.0125, ANOVA — A 2-sided P value less than 0.05 was considered statistically significant. However, the significance level (α) was adjusted to 0.0125 to account for multiple testing; Mean Difference (Final Values) = 3.77, 95% CI 2-sided [3.15 to 4.39] — The main analysis was based on LOCF for missing value

2. Primary Outcome: Prealbumin
Description: Changes in blood prealbumin levels
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Self Control
Number analyzed (Participants) | 142
mg/L | 44.23 (81.77)
Statistical Analysis 1: Comparison: Self Control; Test type: Superiority — >60 mg/L change in prealbumin from baseline to month 6; p = 0.0125, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 39.77, 95% CI 2-sided [26.66 to 56.87] — The main analysis was based on LOCF for missing value

ADVERSE EVENTS:
Time Frame: From the beginning to the end of the study, the time span is from December 2023 to January 2025.Follow up with each subject for 6 months and record adverse events
Groups:
- Adverse Event: Adverse Event (AE) refers to any harmful medical event that occurs during a clinical trial, regardless of whether it is causally related to the investigational drug. Adverse events include the following situations:
  Adverse Reaction (AR) related to the investigational drug: refers to any harmful medical event caused by the pharmacological effects or other reasons of the investigational drug under normal usage conditions.
  Adverse events unrelated to the investigational drug: Refers to any harmful medical event that occurs during a clinical trial, but is scientifically determined to have no causal relationship with the investigational drug.
  Serious Adverse Event (SAE): refers to any harmful medical event that occurs during a clinical trial, regardless of whether it is causally related to the investigational drug, resulting in one of the following consequences:
  Causing death; Endangering life (i.e., if not intervened in a timely manner, it may lead to death); Need for hospitalization or extended hospitalization; Causing persistent or significant disability or functional impairment; Causing congenital malformations or birth defects; Significant medical interventions (such as surgery, blood transfusions, etc.) are required.
Arm/Group | Adverse Event
All-Cause Mortality (participants affected / at risk) | 1/149
Serious Adverse Events (participants affected / at risk) | 31/149
Other Adverse Events (participants affected / at risk) | 3/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Event (N=149)
Peritonitis (Infections and infestations) | 17
Diabetic foot infection (Infections and infestations) | 4
Respiratory system infection (Respiratory, thoracic and mediastinal disorders) | 3
Inguinal hernia (Surgical and medical procedures) | 3
Gastrointestinal lesions and fatigue (Gastrointestinal disorders) | 2
Subcutaneous tunnel infection (Infections and infestations) | 1
Displacement of peritoneal dialysis catheter (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.67% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Event (N=149)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Allergic reaction (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT06358820/Prot_SAP_000.pdf